CLINICAL TRIAL: NCT05500690
Title: Understanding Effects of Folic Acid on the Methylosome and Transcriptome of Women With Spina Bifida Affected Pregnancies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Neurosciences and Hospital, Dhaka (Other Government)
Responsible Party: Principal Investigator, Maitreyi Mazumdar, Associate Professor of Neurology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-P00043006
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy; Spina Bifida, Fetal; Environmental Exposure
Keywords: Spina Bifida; Folic Acid; DNA Methylation; arsenic
MeSH Terms: conditions — Spinal Dysraphism | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Folic Acid (Experimental): 5 mg folic acid supplement by mouth once a day for 12 weeks
  Interventions: Dietary Supplement: Folic Acid Tablet

INTERVENTIONS:
Dietary Supplement: Folic Acid Tablet — 5 mg folic acid supplement

SUMMARY:
Folic acid is currently considered to be the standard of care for primary and secondary prevention of spina bifida, but the mechanisms underlying folic acid's benefits are unknown. One hypothesis is that folic acid changes DNA methylation and transcription of genes important in neural tube closure.

In this study, the investigators will evaluate how DNA methylation of genes associated with neural tube closure changes after a short course of standard-of-care folic acid supplementation. In addition, the investigators will assess whether environmental arsenic exposure modifies the effects of folic acid on the methylosome.

DETAILED DESCRIPTION:
The investigators will encourage women who have recently had a pregnancy affected by spina bifida to take daily folic acid supplements for three months. Folic acid supplementation is considered standard of care for primary and secondary prevention of spina bifida. The investigators will compare DNA methylation in blood and folate levels before and after folic acid use.

ELIGIBILITY:
Inclusion Criteria:

* Women (18+) with a prior pregnancy affected by spina bifida
* Available for required study visits

Exclusion Criteria:

* Personal history of diabetes or gestational diabetes
* Current anticonvulsant medication use
* History of pregnancy affected by identified genetic syndrome associated with neural tube defect such as Trisomy 18
* Current pregnancy
* Abnormal peripheral blood film results (suggestive of megaloblastic anemia/B12 deficiency.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes in DNA Methylation patterns | Week 1 and Week 12
  The investigators will use DNA methylation arrays to compare methylation patterns before and after course of folic acid.

SECONDARY OUTCOMES:
Changes in serum folate concentration | Week 1 and Week 12
  Chemiluminescent Microparticle Immunoassay will be used to measure folate concentration. The investigators will assess changes in serum folate concentration before and after folic acid use.

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Mazumdar, MD, MPH, Principal Investigator — Boston Children's Hospital; Sudipta K Mukherjee, MBBS, MS, Principal Investigator — National Institute of Neurosciences and Hospital, Dhaka
Locations (1):
- National Institute of Neurosciences and Hospital, Dhaka, Bangladesh